CLINICAL TRIAL: NCT01705782
Title: Metabolic Effects of Endotoxin Induced Acute Inflammation in Healthy Young Men With and Without Supplement of Amino Acids.
Brief Title: The Effects of Amino Acid Supplement During Acute Inflammation.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Nikolaj Fibiger Rittig, MD (medical graduate) and Ph.d.-student, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2012-410-12
Record Dates: First submitted 2012-10-08; First posted 2012-10-12 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Febrile Illness Acute; Inflammation; Metabolic Diseases
MeSH Terms: conditions — Inflammation; Metabolic Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Saline (No Intervention): Only saline is given.
- + Saline (Placebo Comparator): Endotoxin is given + Placebo (Saline)
  Interventions: Biological: E. coli endotoxin, US standard
- + amino acids (Active Comparator): Endotoxin is given + amino acids (intravenously)
  Interventions: Biological: E. coli endotoxin, US standard

INTERVENTIONS:
Biological: E. coli endotoxin, US standard
  Arms: + Saline; + amino acids

SUMMARY:
The purpose of the study is to investigate the metabolic effects during acute inflammation with and without the nutritional supplement of amino acids.

E. Coli Endotoxin (LPS, lipopolysaccharide) is used to initiate an inflammatory response.

The study is an interventional randomized placebo study including 8 healthy male subjects. Each subject participates 3 times (different days) and are given one of following interventions:

* Placebo (NaCl)
* Endotoxin, US standard reference E.Coli + Placebo (NaCl)
* Endotoxin, US standard reference E.Coli + Amino acids (intravenously)

It is our hypothesis that the nutritional intervention during acute inflammation plays an important role in lipid and protein metabolism.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* 20<BMI<30
* Age > 25 years old
* Written consent before starting the study

Exclusion Criteria:

* Allergy for soya products ore egg
* Diabetes
* Epilepsy
* Infection
* Immune defects
* Heart disease
* Dysregulated hypertension
* Participating in other trials using radioactive tracers or x-rays the last year.

Min Age: 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-10; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Protein catabolism during acute illness | After 6 hours intervention
  Protein catabolism is measured with amino acid tracer techniques comparing radioactive marked amino acids from blood samples.

SECONDARY OUTCOMES:
The local effects on muscle and fat tissue | At 2 hours and 4,5 hours
  A muscle + fat biopsy are taken twice during the intervention to focus on the local effects in these tissues.
Other systemic metabolic effects during acute illness | 6 hours
  Lipid and glucose metabolism are measured with tracer techniques with radioactive marked glucose + lipid.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical Department MEA, NBG, Aarhus University Hospital, Aarhus C, Jylland, Denmark

REFERENCES:
- [Derived] Pedersen MGB, Lauritzen ES, Svart MV, Stoy J, Sondergaard E, Thomsen HH, Kampmann U, Bjerre M, Jessen N, Moller N, Rittig N. Nutrient sensing: LEAP2 concentration in response to fasting, glucose, lactate, and beta-hydroxybutyrate in healthy young males. Am J Clin Nutr. 2023 Dec;118(6):1091-1098. doi: 10.1016/j.ajcnut.2023.10.007. Epub 2023 Oct 14. PMID 37844838
- [Derived] Vladimirova YV, Molmer MK, Antonsen KW, Moller N, Rittig N, Nielsen MC, Moller HJ. A New Serum Macrophage Checkpoint Biomarker for Innate Immunotherapy: Soluble Signal-Regulatory Protein Alpha (sSIRPalpha). Biomolecules. 2022 Jul 4;12(7):937. doi: 10.3390/biom12070937. PMID 35883493
- [Derived] Rittig N, Bach E, Thomsen HH, Pedersen SB, Nielsen TS, Jorgensen JO, Jessen N, Moller N. Regulation of Lipolysis and Adipose Tissue Signaling during Acute Endotoxin-Induced Inflammation: A Human Randomized Crossover Trial. PLoS One. 2016 Sep 14;11(9):e0162167. doi: 10.1371/journal.pone.0162167. eCollection 2016. PMID 27627109
- [Derived] Rittig N, Bach E, Thomsen HH, Johannsen M, Jorgensen JO, Richelsen B, Jessen N, Moller N. Amino acid supplementation is anabolic during the acute phase of endotoxin-induced inflammation: A human randomized crossover trial. Clin Nutr. 2016 Apr;35(2):322-330. doi: 10.1016/j.clnu.2015.03.021. Epub 2015 Apr 9. PMID 25896101